CLINICAL TRIAL: NCT05008406
Title: E-Learning During COVID-19 Pandemic: Turning a Crisis Into Opportunity
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Amjad Bani Hani, Associate professor, University of Jordan
Other Study IDs: 2020/8
Record Dates: First submitted 2021-07-22; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Satisfaction
MeSH Terms: conditions — Personal Satisfaction | interventions — Physician Engagement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preclinical medical students
  Interventions: Other: Satisfaction
- Clinical medical students
  Interventions: Other: Satisfaction

INTERVENTIONS:
Other: Satisfaction — Students Satisfaction

SUMMARY:
E-learning is now a well-established method of education all over the world, and it has been used for years as a major method of teaching in many fields. The medical field is not far away, but the use of e-learning in it has become increasing, and the technological advances have made this process more realistic and interactive.

The emergence and spread of COVID-19 virus as a global pandemic has placed many restrictions on daily life activities including enrolment in schools and universities in many countries, including Jordan, which has led to a marked and increased use of e-learning as a significant alternative to traditional education. Medical teaching has some peculiar characteristics, especially the need for direct interaction between the student and the patient, attending clinics, wards, and operating rooms, and the close exposure to clinical cases. This have created some restrictions and obstacles in the way of using e-learning in medicine education, in addition to other important influencing and limiting barriers, such as technical barriers, especially in the light of the abrupt transition to e-learning utilization under the current circumstance, and the psychological barriers -in terms of anxiety and stress- that resulted by this pandemic and the consequent home quarantine.

This cross-sectional study aims to study the current state of e-learning in the School of Medicine at the University of Jordan, by evaluating the teaching tools used and the effect of the rapid transition in basic medical teaching and clinical medical training to become mainly based on the e-learning methodology on the academic achievement and assimilation of the clinical part of the medical courses, and the general satisfaction of the medical students at their different academic levels. Other influencing factors will be studied, such as the extent of students' readiness and preparedness to use the e-learning tools and their previous experience in it, the extent of the readiness and experience of their teachers, and the general mental health status of students and their effects on accepting the distance e-learning process, and the commitment to participate and interact with various electronic activities.

This study, after exploring the difficulties and hurdles facing the e-learning process and after analysis, aims to propose practical solutions to facilitate and maintain it beyond the COVID-19 pandemic era.

ELIGIBILITY:
Inclusion Criteria:

* All Medical Students

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Medical Students at The school of medicine at The University of Jordan
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Student's satisfaction Assessed by Lickert scale | 3 months
  Percentage of Students satisfied with distant learning

CONTACTS AND LOCATIONS:
Overall Officials: Amjad Bani Hani, MD, Principal Investigator — The University of Jordan
Locations (1):
- The University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No